CLINICAL TRIAL: NCT01161394
Title: Effect of Pioglitazone on Oxidative Load, Inflammatory End-Points and Vascular Reactivity in Obese Non-Diabetic Patients: A Dose Ranging Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University at Buffalo (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Principal Investigator, Paresh Dandona, Principal Investigator, University at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1851
Record Dates: First submitted 2010-07-12; First posted 2010-07-13 (Estimated); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pioglitazone 15mg (Experimental): 8 patient will receive this drug
  Interventions: Drug: Pioglitazone 15mg
- pioglitazone 30mg (Experimental): 8 patients will get this drug
  Interventions: Drug: pioglitazone 30mg
- Placebo (Placebo Comparator): 8 patient will get this drug
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Pioglitazone 15mg
  Arms: Pioglitazone 15mg
Drug: pioglitazone 30mg
  Arms: pioglitazone 30mg
Drug: placebo
  Arms: Placebo

SUMMARY:
Pioglitazone decreases oxidative load, inflammatory end points and improves vascular reactivity in obese patients in a dose dependent manner and that this effect is independent of its glucose lowering effects.

DETAILED DESCRIPTION:
This is a single center, open labeled study. A total of 24 obese patients will be recruited to participate in this study. The study will have three groups of 8 patients each. Subjects will be enrolled into each group by alternate recruitment. Subjects in group one will receive 15mg of pioglitazone; subjects in group two will receive 30 mg of pioglitazone; subjects in group three will receive placebo. All subjects will receive Pioglitazone or placebo for 6 weeks, followed by a 6-week observation period off Pioglitazone/placebo.

At baseline, and at week 1, week 2, week 4, week 6 and month 3 all patients will have blood drawn for TBARS, ortho and meta-tyrosine, 9-HODE and 13-HODE, NF, Ikb, TNF-a, ICAM-1, VCAM-1, PAI-1, AP-1, EGR-1, MMP-2, MMP-9, TIMP, CRP-1, E-Selectin, P-Selectin, Asymmetric dimethylarginine (ADMA), PAPP-A, SAA, MCP-1, IL-6, ROS generation, insulin levels, and CRP.

Post-ischemic dilation of the brachial artery will be used as an index of endothelium-mediated vasodilation. All subjects will have an oral glucose tolerance test (GTT) with 75gm of glucose at Day 0 and at Day 42. Vascular reactivity will be assessed at 0, 6, and at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* • Obese (BMI>=30)

  * Age: 20 to 65 years of age inclusive
  * Without established clinical coronary artery disease (documented history or myocardial infarction, typical angina and an exercise ECG positive for ischemia or angiographic evidence of CAD)
  * Good health as evidence by History and Physical exam
  * Female subjects must be:

Postmenopausal for at least one year or Surgically incapable of childbearing (i.e. have had a hysterectomy or tubal ligation) or, if capable of childbearing a subject, must be practicing an acceptable method of contraception.

• Subject will be available for duration of the study and willing to comply with all study requirements.

Exclusion Criteria:

* • Diabetes Mellitus

  * Allergy or sensitivity to Pioglitazone
  * Current use of Insulin therapy.
  * Coronary event or procedure (myocardial infarction, unstable angina, coronary artery bypass, surgery or coronary angioplasty) in the previous four weeks
  * Hepatic disease (transaminase > 3 times normal)
  * Renal impairment (Creatinine clearance < 50 mL/min)
  * History of drug or alcohol abuse
  * COPD
  * Participation in any other concurrent clinical trial
  * Any other life-threatening, non-cardiac disease
  * Use of an investigational agent or therapeutic regimen within 30 days of study
  * Pregnancy or nursing

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Inflammation | 12 weeks
  Percent change in NFkb at baseline and after 1, 2, 4, 6, and 12 weeks of pioglitazone therapy.

SECONDARY OUTCOMES:
inflammation | 12 weeks
  TBARS (Thiobarbituric acid reactive substances), ortho and meta-tyrosine, 9-HODE and 13-HODE (hydroxyoctadecadieonic acid derivatives), Cellular/nuclear fractions and DNA binding activity of Nuclear Factor kb, Ikb (inhibitory kappa B), TNF-a(Tumor necrosis factor a), ICAM-1 (Intracellular adhesion molecule 1), VCAM-1(Vascular adhesion molecule 1), PAI-1 (Plasminogen Activator Inhibitor -1) and CRP (C-Reactive protein) and %change in vascular reactivity.

CONTACTS AND LOCATIONS:
Overall Officials: Paresh Dandona, MD, Principal Investigator — Kaleida Health
Locations (1):
- Millard Fillmore gates Hospital, Buffalo, New York, United States